CLINICAL TRIAL: NCT04042350
Title: A Retrospective Analysis Assessing Clinical Risk Factors for Cardiovascular Events and Mortality and Development of a Risk Calculator in Chronic Kidney Disease Stage 5 on Dialysis Treatment Using Data From the AURORA Study
Brief Title: Retrospective Analysis Assessing Clinical Risk Factors for Cardiovascular Events and Mortality and Development of a Risk Calculator in Chronic Kidney Disease Stage 5 on Dialysis
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 1517-MA-3256
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: AURORA; Cardiovascular Events; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CKD patients on dialysis: Data will be analyzed from CKD patients on dialysis that participated in the AURORA study.
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Exploring clinical risk factors associated with the risk for cardiovascular events and mortality, rather than to evaluate specific drugs.

SUMMARY:
The purpose of this study is to evaluate which clinical and laboratory factors are associated with major adverse cardiovascular event (MACE) in chronic kidney disease (CKD) patients on dialysis.

The study will also establish a cardiovascular (CV) risk equation appropriate for this dialysis population.

DETAILED DESCRIPTION:
This study is a retrospective analysis of dialysis dependent CKD patients participating in AURORA. The retrospective analysis will be performed using the AURORA study database.

AURORA was a prospective clinical trial in which dialysis patients were randomly assigned to rosuvastatin or placebo, sponsored by AstraZeneca. Patients included in the AURORA study who had end stage renal disease (ESRD) and had been treated with regular hemodialysis or hemofiltration for at least 3 months. Patients were recruited from approximately 300 centers in 25 countries.

The clinical study data is held by AstraZeneca AB, Sweden.

No formal sample size calculation was performed. The sample size is based on the available data from the AURORA study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in the AURORA study. In brief, men and women who had ESRD and had been treated with regular hemodialysis or hemofiltration for at least 3 months (patients were recruited from 280 centers in 25 countries).

Exclusion Criteria:

* The major exclusion criteria in AURORA were statin therapy within the previous 6 months, expected kidney transplantation within 1 year, and serious hematologic, neoplastic, gastrointestinal, infectious, or metabolic disease (excluding diabetes) that was predicted to limit life expectancy to less than 1 year.
* Other exclusion criteria were a history of a malignant condition, active liver disease (indicated by an alanine aminotransferase level that was more than three times the upper limit of the normal range), uncontrolled hypothyroidism, and an unexplained elevation in the creatine kinase level to more than three times the upper limit of the normal range.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the AURORA study were men and women who had ESRD and had been treated with regular hemodialysis or hemofiltration for at least 3 months.
Sampling Method: Probability Sample
Enrollment: 2773 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Time to first major adverse cardiovascular event (MACE) | Up to a maximum of 5.6 years
  A MACE is defined as a non-fatal myocardial infarction (MI), non-fatal stroke, and CV mortality.

SECONDARY OUTCOMES:
Time to a composite of any CV events | Up to a maximum of 5.6 years
  CV events include non-fatal MI, unstable angina, coronary revascularization therapy, new onset heart failure, non-fatal stroke or all-cause mortality.
Time to CV event: MI | Up to a maximum of 5.6 years
  Time to individual CV event.
Time to CV event: stroke (ischemic or hemorrhagic) | Up to a maximum of 5.6 years
  Time to individual CV event.
Time to CV event: unstable angina | Up to a maximum of 5.6 years
  Time to individual CV event.
Time to CV event: coronary revascularization therapy | Up to a maximum of 5.6 years
  Time to individual CV event.
Time to CV event: new onset heart failure | Up to a maximum of 5.6 years
  Time to individual CV event.
Time to CV mortality | Up to a maximum of 5.6 years
  Time to death caused by a CV event.
Time to all-cause mortality | Up to a maximum of 5.6 years
  Time to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Europe Ltd.
Locations (1):
- Site SE46001, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=377